CLINICAL TRIAL: NCT03150862
Title: A Phase 1b/2 Study to Assess the Safety, Tolerability and Efficacy of BGB-290 in Combination With Radiation Therapy (RT) and/or Temozolomide (TMZ) in Subjects With First-line or Recurrent/Refractory Glioblastoma
Brief Title: A Study Assessing Pamiparib With Radiation and/or Temozolomide (TMZ) in Participants With Newly Diagnosed or Recurrent Glioblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BeiGene USA, Inc. (Industry)
Responsible Party: Sponsor
Organization: BeiGene (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-290-104; 2017-001554-33 (EudraCT Number)
Record Dates: First submitted 2017-05-08; First posted 2017-05-12 (Actual); Results first posted 2022-05-31 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2022-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: Adult glioblastoma, adult giant cell glioblastoma, adult gliosarcoma, glioma neoplasms; recurrent adult brain tumor; neoplasms, central nervous system neoplasms, neoplasms by histologic type, neoplasms by site; astrocytoma; neuroepithelial; neuroectodermal tumors; germ cell and embryonal; antineoplastic agents; glandular and epithelial; nerve tissue, nervous system diseases; temozolomide; BGB-290; alkylating, alkylating agents; molecular mechanisms of pharmacological action; Poly(ADP-ribose) polymerase inhibitors; enzyme inhibitors
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma; Brain Neoplasms; Neoplasms; Neoplasms by Histologic Type; Neoplasms by Site; Astrocytoma; Neuroectodermal Tumors; Nervous System Diseases | interventions — pamiparib; Radiation

STUDY DESIGN:
Masking Description: No Masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A (Dose Escalation) (Experimental): Participants with newly diagnosed unmethylated GBM will receive Pamiparib and radiation therapy.
  Interventions: Drug: Pamiparib; Radiation: Radiation
- Arm B (Dose Escalation) (Experimental): Participants with newly diagnosed unmethylated GBM will receive Pamiparib, radiation therapy (RT) and temozolomide (TMZ).
  Interventions: Drug: Pamiparib; Drug: TMZ; Radiation: Radiation
- Arm A (Dose Expansion) (Experimental): Participants with newly diagnosed unmethylated GBM will receive Pamiparib and radiation therapy.
  Interventions: Drug: Pamiparib; Radiation: Radiation
- Arm C (Dose Escalation) (Experimental): Participants with recurrent/refractory methylated or unmethylated GBM will receive Pamiparib and TMZ.
  Interventions: Drug: Pamiparib; Drug: TMZ
- Arm C (Dose Expansion-Cohorts C1 and C2) (Experimental): Participants with recurrent/refractory methylated or unmethylated GBM will receive Pamiparib and TMZ.
  Interventions: Drug: Pamiparib; Drug: TMZ

INTERVENTIONS:
Drug: Pamiparib — Administered as specified in the treatment arm
  Other Names: BGB-290
Drug: TMZ — Administered as specified in the treatment arm
  Arms: Arm B (Dose Escalation); Arm C (Dose Escalation); Arm C (Dose Expansion-Cohorts C1 and C2)
Radiation: Radiation — Up to 60 Gy (total) over 6 - 7 weeks
  Arms: Arm A (Dose Escalation); Arm A (Dose Expansion); Arm B (Dose Escalation)

SUMMARY:
The primary objective of this study is to evaluate the safety, efficacy and clinical activity of Pamiparib in combination with radiation therapy (RT) and/or temozolomide (TMZ) in participants with newly diagnosed or recurrent/refractory glioblastoma.

DETAILED DESCRIPTION:
An open-label, multiple-dose, dose-escalation study to determine the safety, pharmacokinetics (PK) and pharmacodynamics (PD) of Pamiparib in combination with radiation therapy (RT) and/or TMZ.

In dose escalation/Phase 1b, Pamiparib will be combined with RT (Arm A) or RT and TMZ (Arm B) in participants with newly diagnosed unmethylated glioblastoma (GBM) and in Arm C of the study Pamiparib will be combined with TMZ in participants with methylated or unmethylated recurrent/refractory GBM.

The dose expansion/Phase 2 phase will enroll up to 4 cohorts: participants with newly diagnosed unmethylated GBM in Arms A and B, and 2 cohorts of participants with recurrent/refractory GBM grouped by O-6-methylguanine-DNA methyltransferase (MGMT) status - unmethylated or methylated - in Arm C.

Participants in Arms A and B are treated until completion of RT and participants in Arm C may continue treatment in the absence of safety concerns and disease progression.

ELIGIBILITY:
Key Inclusion Criteria: All participants

1. Age ≥ 18 years old.
2. Confirmed diagnosis of glioblastoma (WHO Grade IV).
3. Agreement to provide archival tumor tissue for exploratory biomarker analysis
4. Ability to undergo serial MRIs.
5. Eastern Cooperative Oncology Group (ECOG) status ≤ 1.
6. Adequate hematologic and end-organ function
7. Females of childbearing potential and non-sterile males must agree to use highly effective methods of birth control throughout the course of study and at least up to 6 months after last dosing.
8. Ability to swallow whole capsules.

   Participants in Arms A and B (not Arm C) must meet inclusion criteria # 9 - 11:
9. No previous treatment for GBM except surgery.
10. Able to start radiation therapy ≤ 49 days after surgery but ≥ 14 days after a biopsy or ≥28 days after an open biopsy or craniotomy with adequate wound healing.
11. Documented unmethylated MGMT promoter status.

    Participants in Arm C Escalation (Phase 1b) must meet inclusion criteria # 12 - 15:
12. Documentation of MGMT promoter status
13. No prior systemic chemotherapy other than TMZ for GBM.
14. Histologically confirmed secondary glioblastoma
15. Disease that is evaluable or measurable as defined by Response Assessment in Neuro-Oncology (RANO) criteria

    Participants in Arm C Expansion (Phase 2), must meet criteria # 16 - 18:
16. Histologically confirmed de novo (primary) glioblastoma with unequivocal first progressive disease (PD) after RT with concurrent/adjuvant TMZ chemotherapy
17. Disease that is measurable as defined by RANO criteria
18. Documentation of MGMT promoter status

Key Exclusion Criteria: All participants

1. Prior chemotherapy, biologic therapy, immunotherapy or investigational agents ≤21 days prior to start of study treatment.
2. Toxicity of ≥ Grade 2 from prior therapy.
3. Major surgery or significant other injury ≤ 4 weeks prior to start of study treatment.
4. History of other active malignancies within 2 years with exception of (i) adequately treated in situ cancer of the cervix, (ii) non-melanoma skin cancer, or (iii) localized adequately treated cancer with curative intent or malignancy diagnosed > 2 years ago with no evidence of disease and no treatment ≤ 2 years prior to study treatment.
5. Active infection requiring systemic treatment.
6. Known human immunodeficiency virus (HIV) or active viral hepatitis.
7. Active, clinically significant cardiac disease or any Class 3 or 4 cardiac disease, ventricular arrhythmia or Cerebrovascular Accident (CVA) ≤ 6 months prior to start of treatment.
8. Active clinically significant gastrointestinal disease.
9. Active bleeding disorder ≤ 6 months prior to start of treatment.
10. Need for therapeutic anti-coagulation with heparin, warfarin or other anticoagulants.
11. Use of any medications or food known to be strong or moderate cytochrome P450, family 3, subfamily A (CYP3A) inhibitors or strong inducers.
12. Pregnant or nursing females.
13. Significant intercurrent illness that may result in participant's death prior to death from glioblastoma.

    Arms B and C Only:
14. Known hypersensitivity to any component of TMZ or decarbazine (DTIC).
15. Have hereditary problems of galactose intolerance

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (22):
- United States (18):
  - Center For Neurosciences, Tucson, Arizona
  - UCLA, Los Angeles, California
  - University of California At San Francisco, San Francisco, California
  - Sarah Cannon Research Institute (Scri) At Health One, Denver, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Midamerica Division, Inc, Kansas City, Missouri
  - Washington University in St Louis, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center Mskcc, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Sarah Cannon Research Institute (Scri) Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University Hospital Jefferson Health, Philadelphia, Pennsylvania
  - Tennessee Oncology, Pllc Nashville, Nashville, Tennessee
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
- Liverpool Hospital, Liverpool, New South Wales, Australia
- Institut Gustave Roussy, Villejuif, France
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- University of Zurich Medical School, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Xiong Y, Guo Y, Liu Y, Wang H, Gong W, Liu Y, Wang X, Gao Y, Yu F, Su D, Wang F, Zhu Y, Zhao Y, Wu Y, Qin Z, Sun X, Ren B, Jiang B, Jin W, Shen Z, Tang Z, Song X, Wang L, Liu X, Zhou C, Jiang B. Pamiparib is a potent and selective PARP inhibitor with unique potential for the treatment of brain tumor. Neoplasia. 2020 Sep;22(9):431-440. doi: 10.1016/j.neo.2020.06.009. Epub 2020 Jul 8. PMID 32652442

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of a dose escalation phase and a dose expansion phase. A total of 116 participants were recruited in Netherlands, Switzerland and United States.
Groups:
- Arm A: Dose Escalation (DE) - Pamiparib 2 Weeks (Wks) + Radiation Therapy (RT) 6 Wks: Participants with newly diagnosed unmethylated glioblastoma (GBM) received 60 milligrams (mg) pamiparib orally twice daily (BID) for 2 weeks in combination with up to 60 Gy radiation for 6 weeks
- Arm A: DE-Pamiparib 4 Wks + RT 6 Wks: Participants with newly diagnosed unmethylated GBM received 60 mg pamiparib orally for 4 weeks in combination with up to 60 Gy radiation for 6 weeks
- Arm A: DE- Pamiparib 6Wks + RT 6 Wks; Arm A: Dose Expansion (E) - Pamiparib 6 Wks + RT 6 Wks: Participants with newly diagnosed unmethylated GBM received 60 mg pamiparib orally for 6 weeks in combination with up to 60 Gy radiation for 6 weeks
- Arm B: DE-Pamiparib 6 Wks + RT 6 Wks + Temozolomide: Participants with newly diagnosed unmethylated GBM received 60 mg pamiparib orally for 6 weeks in combination with up to 60 Gy radiation for 6 weeks and 60 mg temozolomide Wks 1 and 5
- Arm C: DE - Pamiparib + Temozolomide 20 mg: Participants with both methylated and unmethylated recurrent/refractory GBM received 60 mg pamiparib BID and 20 mg temozolomide once daily orally from Day 1 to Day 21
- Arm C: DE - Pamiparib + Temozolomide 40 mg: Participants with both methylated and unmethylated recurrent/refractory GBM received 60 mg pamiparib BID and 40 mg temozolomide once daily orally from Day 1 to Day 21
- Arm C: E- Pamiparib + Temozolomide 60 mg: Participants with both methylated and unmethylated recurrent/refractory GBM received 60 mg pamiparib BID and 60 mg temozolomide once daily orally from Day 1 to Day 7
Period: Overall Study
Arm/Group | Arm A: Dose Escalation (DE) - Pamiparib 2 Weeks (Wks) + Radiation Therapy (RT) 6 Wks | Arm A: DE-Pamiparib 4 Wks + RT 6 Wks | Arm A: DE- Pamiparib 6Wks + RT 6 Wks | Arm A: Dose Expansion (E) - Pamiparib 6 Wks + RT 6 Wks | Arm B: DE-Pamiparib 6 Wks + RT 6 Wks + Temozolomide | Arm C: DE - Pamiparib + Temozolomide 20 mg | Arm C: DE - Pamiparib + Temozolomide 40 mg | Arm C: E- Pamiparib + Temozolomide 60 mg
Started | 3 | 8 | 9 | 40 | 9 | 9 | 8 | 30
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 8 | 9 | 40 | 9 | 9 | 8 | 30
Not completed — Death | 2 | 7 | 8 | 27 | 4 | 8 | 6 | 21
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 3 | 1 | 1 | 1 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Not completed — Sponsor's decision | 0 | 0 | 0 | 10 | 3 | 0 | 1 | 1
Not completed — Change in Methylation status | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Roll over in to Long Term Extension | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set includes all participants who received any study treatment (pamiparib, RT, and/or TMZ). The Safety Analysis Set was used for all efficacy and safety analyses.
Groups:
- Arm A: DE - Pamiparib 2 Wks + Radiation Therapy (RT) 6 Wks: Participants with newly diagnosed unmethylated glioblastoma (GBM) received 60 mg pamiparib orally BID for 2 weeks in combination with up to 60 Gy radiation for 6 weeks
- Total: Total of all reporting groups
Arm/Group | Arm A: DE - Pamiparib 2 Wks + Radiation Therapy (RT) 6 Wks | Arm A: DE-Pamiparib 4 Wks + RT 6 Wks | Arm A: DE- Pamiparib 6Wks + RT 6 Wks | Arm A: Dose Expansion (E) - Pamiparib 6 Wks + RT 6 Wks | Arm B: DE-Pamiparib 6 Wks + RT 6 Wks + Temozolomide | Arm C: DE - Pamiparib + Temozolomide 20 mg | Arm C: DE - Pamiparib + Temozolomide 40 mg | Arm C: E- Pamiparib + Temozolomide 60 mg | Total
Number analyzed (Participants) | 3 | 8 | 9 | 40 | 9 | 9 | 8 | 30 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (8.39) | 63.4 (8.80) | 58.8 (7.66) | 56.7 (13.48) | 60.9 (9.94) | 49.2 (12.63) | 49.1 (15.51) | 58.6 (10.54) | 57.10 (12.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 17 | 4 | 1 | 4 | 10 | 39
  Male | 3 | 7 | 7 | 23 | 5 | 8 | 4 | 20 | 77
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Black or African American | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 3
  White | 3 | 7 | 7 | 38 | 9 | 7 | 8 | 27 | 106
  Unknown/Not Reported | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b Escalation Phase: Number of Participants With Dose-Limiting Toxicities (DLTs) as Assessed by CTCAE
Description: A DLT is defined as one of the following toxicities occurring during the DLT assessment window:
  Grade ≥3 non-hematologic, non-hepatic major organ adverse event (AE) Grade 4 neutropenia lasting >7 days Grade ≥3 febrile neutropenia Grade 3 thrombocytopenia with clinically significant bleeding Grade 4 thrombocytopenia lasting > 3 days and requiring transfusion, or any decreased platelet count <15,000/mm3/ <15.0 x 109/L Grade ≥4 anemia Grade ≥3 total bilirubin or hepatic transaminases (ALT or AST)
Time Frame: Arm A:Day 1 Pamiparib dose until 4 weeks after the last RT; Arm B: Day 1 of Pamiparib and Temozolomide until 4 weeks after the last RT; Arm C: 1st cycle of 28 days
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Arm A: DE - Pamiparib 2 Wks + Radiation Therapy (RT) 6 Wks | Arm A: DE-Pamiparib 4 Wks + RT 6 Wks | Arm A: DE- Pamiparib 6Wks + RT 6 Wks | Arm B: DE-Pamiparib 6 Wks + RT 6 Wks + Temozolomide | Arm C: DE - Pamiparib + Temozolomide 20 mg | Arm C: DE - Pamiparib + Temozolomide 40 mg
Number analyzed (Participants) | 3 | 8 | 9 | 9 | 9 | 8
participants | 0 | 0 | 2 | 1 | 0 | 3

2. Primary Outcome: Phase 1b Escalation Phase: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) as Assessed by CTCAE
Description: A treatment-emergent adverse event (TEAE) is defined as an AE that had an onset date on or after first dose of study treatment or was worsening in severity from baseline (pretreatment) up to 30 days following permanent study treatment discontinuation or initiation of new anti-cancer therapy, whichever occurs first.
  An SAE is any untoward medical occurrence that, at any dose meets at least one of the following criteria: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, is considered a significant medical AE based on medical judgment.
Time Frame: From initiation of study treatment (for TEAE) or from the date informed consent has been signed (for SAE), until 30 days after last study treatment or initiation of new anticancer therapy, whichever occurs first (up to 3 years and 7.5 months)
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Arm A: DE - Pamiparib 2 Wks + Radiation Therapy (RT) 6 Wks | Arm A: DE-Pamiparib 4 Wks + RT 6 Wks | Arm A: DE- Pamiparib 6Wks + RT 6 Wks | Arm B: DE-Pamiparib 6 Wks + RT 6 Wks + Temozolomide | Arm C: DE - Pamiparib + Temozolomide 20 mg | Arm C: DE - Pamiparib + Temozolomide 40 mg
Number analyzed (Participants) | 3 | 8 | 9 | 9 | 9 | 8
participants
  Participants with At Least 1 TEAE | 3 | 8 | 9 | 9 | 9 | 8
  TEAE with Grade 3 or Higher | 1 | 3 | 4 | 4 | 5 | 7
  Treatment Emergent SAEs | 0 | 2 | 2 | 2 | 4 | 3
  TEAE Leading to Death | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Phase 1b Escalation Phase Arm C: Number of Participants With Clinically Relevant Changes in Vital Signs and Clinical Laboratory Measurements
Time Frame: From the date of first dose up to end of study (EOS) visit (up to 3 years and 7.5 months)
Population: Safety Analysis Set
Measure: Number; unit: Number of participants
Arm/Group | Arm C: DE - Pamiparib + Temozolomide 20 mg | Arm C: DE - Pamiparib + Temozolomide 40 mg
Number analyzed (Participants) | 9 | 8
Number of participants | 0 | 0

4. Primary Outcome: Phase 2 Arm A: Modified Disease Control Rate (DCR) as Assessed by Response Assessment in Neuro-Oncology (RANO) Criteria
Description: Modified DCR is defined as the percentage of participants with complete response (CR), partial response (PR) or stable disease (SD) per RANO criteria as the response assessment at the end-of-treatment (EOT) visit.
Time Frame: From the date of first dose up to first documentation of disease progression while participant is alive ( up to 3 years and 7.5 months)
Population: The Efficacy Analysis Set (Arm A) includes participants in the Safety Analysis Set who had a tumor assessment at baseline and at End of Treatment unless discontinued treatment or study early due to disease progression or death prior to tumor assessment. Participants with available data were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Dose Expansion (E) - Pamiparib 6 Wks + RT 6 Wks
Number analyzed (Participants) | 32
Percentage of participants | 65.6 [46.8 to 81.4]

5. Primary Outcome: Phase 2 Arm C: Objective Response Rate (ORR) as Assessed Using RANO Criteria
Description: ORR (objective response rate) is defined as percentage of participants with best overall response of CR or PR per RANO criteria (confirmed by a subsequent tumor assessment at least four weeks apart).
Time Frame: From the date of first dose up to first documentation of disease progression while participant is alive (up to 3 years and 7.5 months)
Population: The Efficacy Analysis Set (Arm C) includes participants in the Safety Analysis Set who had measurable disease at baseline and at least one postbaseline tumor assessment unless discontinued treatment or study early due to disease progression or death prior to tumor assessment. Participants with available data were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm C: E- Pamiparib + Temozolomide 60 mg
Number analyzed (Participants) | 28
Percentage of participants | 10.7 [2.3 to 28.2]

6. Primary Outcome: Phase 1b Arm C: Number of Cycles of Treatment Received by Participants
Description: Data shows the number of participants who received treatment for the given number of cycles.
Time Frame: From the date of first dose up to EOS visit ( up to 3 years and 7.5 months)
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Arm C: DE - Pamiparib + Temozolomide 20 mg | Arm C: DE - Pamiparib + Temozolomide 40 mg
Number analyzed (Participants) | 9 | 8
participants
  <1 cycle | 2 | 3
  1 cycle | 4 | 0
  2 cycles | 1 | 2
  3 cycles | 0 | 1
  4 cycles | 1 | 0
  5 cycles | 1 | 0
  6 cycles | 0 | 0
  7 cycles | 0 | 0
  >7 cycles | 0 | 2

7. Primary Outcome: Phase 1b Arm C: Average Dose Intensity of Pamiparib And TMZ Received Per Participant
Description: The average dose intensity per participant = total dose (mg) per participant / duration of treatment (days).
Time Frame: From the date of first dose until EOS visit (up to 3 years and 7.5 months)
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: milligrams/Day
Arm/Group | Arm C: DE - Pamiparib + Temozolomide 20 mg | Arm C: DE - Pamiparib + Temozolomide 40 mg
Number analyzed (Participants) | 9 | 8
milligrams/Day
  Pamiparib | 97.5 (25.41) | 107.6 (14.65)
  TMZ | 13.6 (1.88) | 28.2 (10.80)

8. Secondary Outcome: Phase 1B and Phase 2: Pharmacokinetics: Ctrough of Pamiparib
Time Frame: Pre-dose, 2 hours post dose on Days 1 and 15 of radiation Therapy
Population: The Pharmacokinetic (PK) Analysis Set includes all participants for whom valid pamiparib PK parameters can be estimated. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm A: DE - Pamiparib 2 Wks + Radiation Therapy (RT) 6 Wks | Arm A: DE-Pamiparib 4 Wks + RT 6 Wks | Arm A: DE- Pamiparib 6Wks + RT 6 Wks | Arm A: Dose Expansion (E) - Pamiparib 6 Wks + RT 6 Wks | Arm B: DE-Pamiparib 6 Wks + RT 6 Wks + Temozolomide | Arm C: DE - Pamiparib + Temozolomide 20 mg | Arm C: DE - Pamiparib + Temozolomide 40 mg | Arm C: E- Pamiparib + Temozolomide 60 mg
Number analyzed (Participants) | 3 | 5 | 6 | 35 | 7 | 6 | 6 | 25
ng/mL | 891.3 (444.51) | 1817.0 (1226.53) | 1848.3 (784.38) | 2239.9 (1011.07) | 2134.3 (953.06) | 1893.3 (718.46) | 1550.8 (1422.55) | 1500.2 (943.35)

9. Secondary Outcome: Phase 1b Arm A and Arm B Escalation Phase: Modified Disease Control Rate as Assessed by RANO Criteria
Description: as for outcome 4
Time Frame: From the date of first dose up to first documentation of disease progression while participant is alive (approximately 3 years and 7.5 months)
Population: Efficacy Analysis Set; Participants with available data were included in the analysis
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: DE - Pamiparib 2 Wks + Radiation Therapy (RT) 6 Wks | Arm A: DE-Pamiparib 4 Wks + RT 6 Wks | Arm A: DE- Pamiparib 6Wks + RT 6 Wks | Arm B: DE-Pamiparib 6 Wks + RT 6 Wks + Temozolomide
Number analyzed (Participants) | 3 | 6 | 7 | 5
Percentage of participants | 66.7 [9.4 to 99.2] | 100.0 [54.1 to 100.0] | 42.9 [9.9 to 81.6] | 80.0 [28.4 to 99.5]

10. Secondary Outcome: Phase 1b Escalation Phase Arm C: Disease Control Rate as Assessed by RANO Criteria
Description: DCR is defined as the percentage of participants with best overall response of CR, PR or SD per RANO criteria. CR or PR will be confirmed by a subsequent tumor assessment at least four weeks apart
Time Frame: as for outcome 5
Population: Efficacy Analysis Set; Participants with available data were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Arm C: DE- Pamiparib + Temozolomide 20 mg: Participants with both methylated and unmethylated recurrent/refractory GBM received 60 mg pamiparib BID and 20 mg temozolomide once daily orally from Day 1 to Day 21
Arm/Group | Arm C: DE- Pamiparib + Temozolomide 20 mg | Arm C: DE - Pamiparib + Temozolomide 40 mg
Number analyzed (Participants) | 9 | 7
Percentage of participants | 55.6 [21.2 to 86.3] | 71.4 [29.0 to 96.3]

11. Secondary Outcome: Phase 1b and Phase 2 Arms A and B: ORR as Assessed Using RANO Criteria
Description: ORR is defined as percentage of participants with best overall response of CR or PR per RANO criteria (confirmed by a subsequent tumor assessment at least four weeks apart).
Time Frame: as for outcome 4
Population: Efficacy Evaluable Analysis Set; Participants with available data were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: DE - Pamiparib 2 Wks + Radiation Therapy (RT) 6 Wks | Arm A: DE-Pamiparib 4 Wks + RT 6 Wks | Arm A: DE- Pamiparib 6Wks + RT 6 Wks | Arm A: Dose Expansion (E) - Pamiparib 6 Wks + RT 6 Wks | Arm B: DE-Pamiparib 6 Wks + RT 6 Wks + Temozolomide
Number analyzed (Participants) | 3 | 6 | 7 | 32 | 5
Percentage of participants | 0 [0.0 to 70.8] | 16.7 [0.4 to 64.1] | 0 [0.0 to 41.0] | 3.1 [0.1 to 16.2] | 0 [0.0 to 52.2]

12. Secondary Outcome: Phase 1b and Phase 2 Arms A, B and C: Clinical Benefit Rate as Assessed Using RANO Criteria
Description: Clinical benefit rate (CBR) is defined as the percentage of participants with best overall response of CR, PR or SD ≥ 24 weeks per RANO criteria (confirmed by a subsequent tumor assessment at least four weeks apart).
Time Frame: as for outcome 5
Population: Efficacy Analysis Set; participants with available data were included in the analysis
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: DE - Pamiparib 2 Wks + Radiation Therapy (RT) 6 Wks | Arm A: DE-Pamiparib 4 Wks + RT 6 Wks | Arm A: DE- Pamiparib 6Wks + RT 6 Wks | Arm A: Dose Expansion (E) - Pamiparib 6 Wks + RT 6 Wks | Arm B: DE-Pamiparib 6 Wks + RT 6 Wks + Temozolomide | Arm C: DE - Pamiparib + Temozolomide 20 mg | Arm C: DE - Pamiparib + Temozolomide 40 mg | Arm C: E- Pamiparib + Temozolomide 60 mg
Number analyzed (Participants) | 3 | 6 | 7 | 32 | 5 | 9 | 7 | 28
Percentage of participants | 0 [0.0 to 70.8] | 33.3 [4.3 to 77.7] | 0 [0.0 to 41.0] | 37.6 [21.1 to 56.3] | 40.0 [5.3 to 85.3] | 0 [0.0 to 33.6] | 28.6 [3.7 to 71.0] | 17.9 [6.1 to 36.9]

13. Secondary Outcome: Phase 1b and Phase 2 Arms A, B and C: Duration of Response (DOR) as Assessed Using RANO Criteria
Description: DOR is defined as the time from the date of the earliest documented response to disease progression or death for any cause whichever occurs earlier (confirmed by a subsequent tumor assessment at least four weeks apart).
Time Frame: From first documentation of CR or PR to first documentation of disease progression or death (up to 3 years and 7.5 months)
Population: Efficacy Analysis Set; Only the participants with objective responses were included in DOR analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: DE - Pamiparib 2 Wks + Radiation Therapy (RT) 6 Wks | Arm A: DE-Pamiparib 4 Wks + RT 6 Wks | Arm A: DE- Pamiparib 6Wks + RT 6 Wks | Arm A: Dose Expansion (E) - Pamiparib 6 Wks + RT 6 Wks | Arm B: DE-Pamiparib 6 Wks + RT 6 Wks + Temozolomide | Arm C: DE - Pamiparib + Temozolomide 20 mg | Arm C: DE - Pamiparib + Temozolomide 40 mg | Arm C: E- Pamiparib + Temozolomide 60 mg
Number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3
Months |  | 6.44 [NA to NA] — NA = NE; Not estimable due to insufficient number of events |  | 10.32 [NA to NA] — NA = NE; Not estimable due to insufficient number of events |  |  | 11.7 [NA to NA] — NA = NE; Not estimable due to insufficient number of events | NA [12.68 to NA] — NA = NE; Not estimable due to insufficient number of events

14. Secondary Outcome: Phase 1b and Phase 2 Arms A, B and C: Progression Free Survival (PFS) as Assessed Using RANO Criteria
Description: PFS is defined as the time from the first dose date to disease progression per RANO criteria or death, whichever occurs first.
Time Frame: From the date of first dose up to first documentation of disease progression or death (up to 3 years and 7.5 months)
Population: Safety Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: DE - Pamiparib 2 Wks + Radiation Therapy (RT) 6 Wks | Arm A: DE-Pamiparib 4 Wks + RT 6 Wks | Arm A: DE- Pamiparib 6Wks + RT 6 Wks | Arm A: Dose Expansion (E) - Pamiparib 6 Wks + RT 6 Wks | Arm B: DE-Pamiparib 6 Wks + RT 6 Wks + Temozolomide | Arm C: DE - Pamiparib + Temozolomide 20 mg | Arm C: DE - Pamiparib + Temozolomide 40 mg | Arm C: E- Pamiparib + Temozolomide 60 mg
Number analyzed (Participants) | 3 | 8 | 9 | 40 | 8 | 9 | 8 | 30
Months | 3.12 [2.79 to 3.29] | 8.94 [3.78 to 11.56] | 2.56 [2.14 to NA] — NA = NE; Not estimable to due to insufficient number of events | 4.44 [3.29 to 6.24] | 5.75 [2.37 to 6.47] | 1.81 [0.82 to 3.48] | 2.66 [0.66 to 7.39] | 1.87 [1.48 to 1.91]

15. Secondary Outcome: Phase 1b and Phase 2 Arms A, B and C: Overall Survival (OS)
Description: OS is defined as the time from the first dose date to date of death for any cause.
Time Frame: From the date of first dose up to the date of death (up to 3 years and 7.5 months)
Population: Safety Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: DE - Pamiparib 2 Wks + Radiation Therapy (RT) 6 Wks | Arm A: DE-Pamiparib 4 Wks + RT 6 Wks | Arm A: DE- Pamiparib 6Wks + RT 6 Wks | Arm A: Dose Expansion (E) - Pamiparib 6 Wks + RT 6 Wks | Arm B: DE-Pamiparib 6 Wks + RT 6 Wks + Temozolomide | Arm C: DE - Pamiparib + Temozolomide 20 mg | Arm C: DE - Pamiparib + Temozolomide 40 mg | Arm C: E- Pamiparib + Temozolomide 60 mg
Number analyzed (Participants) | 3 | 8 | 9 | 40 | 8 | 9 | 8 | 30
Months | 14.46 [13.93 to 14.98] | 13.44 [4.14 to 20.24] | 10.25 [4.44 to 19.84] | 12.71 [9.79 to 14.46] | 14.23 [7.98 to NA] — NA = NE; Not estimable due to insufficient number of events | 6.00 [2.60 to 9.79] | 8.62 [2.96 to NA] — NA = NE; Not estimable due to insufficient number of events | 7.79 [6.21 to 10.68]

16. Secondary Outcome: Phase 2 Arms A and C Expansion Phase: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: Safety Analysis Set
Measure: Number; unit: Number of participants
Arm/Group | Arm A: Dose Expansion (E) - Pamiparib 6 Wks + RT 6 Wks | Arm C: E- Pamiparib + Temozolomide 60 mg
Number analyzed (Participants) | 40 | 30
Number of participants
  Participants with at Lease 1 TEAE | 40 | 29
  TEAE with Grade 3 or Higher | 25 | 19
  Treatment Emergent SAEs | 18 | 11
  TEAE Leading to Death | 3 | 1

17. Secondary Outcome: Phase 2 Expansion Phase Arm A and C: Number of Participants With Clinically Relevant Changes in Vital Signs and Clinical Laboratory Measurements
Time Frame: From the date of first dose up to EOS visit (up to 3 years and 7.5 months)
Population: Safety Analysis Set
Measure: Number; unit: Number of participants
Arm/Group | Arm A: Dose Expansion (E) - Pamiparib 6 Wks + RT 6 Wks | Arm C: E- Pamiparib + Temozolomide 60 mg
Number analyzed (Participants) | 40 | 30
Number of participants | 0 | 0

18. Secondary Outcome: Phase 2 Arms A and C Expansion Phase: Number of Cycles of Treatment Received by Participants
Description: Data shows the number of participants who received treatment for the given number of cycles.
Time Frame: From date of first dose up to EOS Visit (up to 3 years and 7.5 months)
Population: Safety Analysis Set; For Arm A Only participants who entered the maintenance phase were included in the analysis as per protocol.
Measure: Number; unit: participants
Arm/Group | Arm A: Dose Expansion (E) - Pamiparib 6 Wks + RT 6 Wks | Arm C: E- Pamiparib + Temozolomide 60 mg
Number analyzed (Participants) | 29 | 30
participants
  <1 cycle | 3 | 8
  1 cycle | 9 | 8
  2 cycles | 2 | 7
  3 cycles | 2 | 1
  4 cycles | 3 | 1
  5 cycles | 3 | 0
  6 cycles | 3 | 0
  7 cycles | 0.0 | 0
  >7 cycles | 4 | 5

19. Secondary Outcome: Phase 2 Arms A and C Expansion Phase: Average Dose Intensity of Pamiparib and TMZ Received Per Participant
Description: The average dose intensity per participant = total dose (mg) per participant / duration of treatment (days).
Time Frame: From date of first dose up to EOS Visit (up to 3 years and 7.5 months)
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: Milligrams/Day
Arm/Group | Arm A: Dose Expansion (E) - Pamiparib 6 Wks + RT 6 Wks | Arm C: E- Pamiparib + Temozolomide 60 mg
Number analyzed (Participants) | 40 | 30
Milligrams/Day
  Pamiparib | 109.0 (22.07) | 109.5 (15.22)
  TMZ | NA (NA) — NA = Not applicable since no TMZ was administered in this arm | 19.6 (11.60)

ADVERSE EVENTS:
Time Frame: From initiation of study treatment (for TEAE) or from the date informed consent has been signed (for SAE), until 30 days after last study treatment or initiation of new anticancer therapy, whichever occurs first (up to 3 years and 7.5 months)
Description: A treatment-emergent adverse event (TEAE) is defined as an AE that had an onset date on or after first dose of study treatment or was worsening in severity from baseline (pretreatment) up to 30 days following permanent study treatment discontinuation or initiation of new anti-cancer therapy, whichever occurs first.
Groups:
- Arm 1Arm A: DE - Pamiparib 2 Wks + Radiation Therapy (RT) 6 Wks: Participants with newly diagnosed unmethylated glioblastoma (GBM) received 60 mg pamiparib orally BID for 2 weeks in combination with up to 60 Gy radiation for 6 weeks
Arm/Group | Arm 1Arm A: DE - Pamiparib 2 Wks + Radiation Therapy (RT) 6 Wks | Arm A: DE-Pamiparib 4 Wks + RT 6 Wks | Arm A: DE- Pamiparib 6Wks + RT 6 Wks | Arm A: Dose Expansion (E) - Pamiparib 6 Wks + RT 6 Wks | Arm B: DE-Pamiparib 6 Wks + RT 6 Wks + Temozolomide | Arm C: DE - Pamiparib + Temozolomide 20 mg | Arm C: DE - Pamiparib + Temozolomide 40 mg | Arm C: E- Pamiparib + Temozolomide 60 mg
All-Cause Mortality (participants affected / at risk) | 2/3 | 7/8 | 8/9 | 27/40 | 4/9 | 8/9 | 6/8 | 21/30
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/8 | 2/9 | 18/40 | 2/9 | 4/9 | 3/8 | 11/30
Other Adverse Events (participants affected / at risk) | 3/3 | 8/8 | 9/9 | 40/40 | 9/9 | 9/9 | 7/8 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1Arm A: DE - Pamiparib 2 Wks + Radiation Therapy (RT) 6 Wks (N=3) | Arm A: DE-Pamiparib 4 Wks + RT 6 Wks (N=8) | Arm A: DE- Pamiparib 6Wks + RT 6 Wks (N=9) | Arm A: Dose Expansion (E) - Pamiparib 6 Wks + RT 6 Wks (N=40) | Arm B: DE-Pamiparib 6 Wks + RT 6 Wks + Temozolomide (N=9) | Arm C: DE - Pamiparib + Temozolomide 20 mg (N=9) | Arm C: DE - Pamiparib + Temozolomide 40 mg (N=8) | Arm C: E- Pamiparib + Temozolomide 60 mg (N=30)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Apraxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral cyst (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemiplegia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychogenic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasogenic cerebral oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1Arm A: DE - Pamiparib 2 Wks + Radiation Therapy (RT) 6 Wks (N=3) | Arm A: DE-Pamiparib 4 Wks + RT 6 Wks (N=8) | Arm A: DE- Pamiparib 6Wks + RT 6 Wks (N=9) | Arm A: Dose Expansion (E) - Pamiparib 6 Wks + RT 6 Wks (N=40) | Arm B: DE-Pamiparib 6 Wks + RT 6 Wks + Temozolomide (N=9) | Arm C: DE - Pamiparib + Temozolomide 20 mg (N=9) | Arm C: DE - Pamiparib + Temozolomide 40 mg (N=8) | Arm C: E- Pamiparib + Temozolomide 60 mg (N=30)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 13 (19) | 4 (7) | 3 (3) | 3 (6) | 6 (15)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 1 (1) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 1 (2) | 3 (3)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema of eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 5 (8) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breath odour (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 14 (16) | 3 (3) | 2 (2) | 2 (2) | 12 (17)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 12 (17) | 2 (2) | 2 (2) | 1 (1) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 5 (5) | 29 (42) | 7 (8) | 4 (4) | 4 (5) | 13 (18)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth discolouration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 13 (20) | 2 (2) | 1 (1) | 4 (5) | 7 (15)
Vomiting projectile (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 2 (2) | 6 (7) | 29 (34) | 6 (7) | 1 (1) | 4 (4) | 17 (20)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 3 (4)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Swelling face (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic lesion (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 5 (6) | 1 (1) | 0 (0) | 3 (3) | 5 (8)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pseudomeningocele (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radiation injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Blood bilirubin unconjugated increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Cortisol decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 3 (3) | 1 (1) | 4 (5)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 6 (9) | 3 (3) | 2 (2) | 2 (2) | 5 (10)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 7 (8) | 1 (2) | 3 (3) | 1 (1) | 8 (18)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 9 (10) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 6 (8) | 4 (7) | 2 (2) | 1 (1) | 6 (10)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3) | 14 (15) | 4 (4) | 2 (2) | 1 (1) | 7 (8)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal hamartoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 6 (7) | 1 (2) | 1 (1) | 0 (0) | 3 (3)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 11 (12) | 2 (2) | 1 (1) | 1 (1) | 8 (8)
Drooling (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 10 (11) | 2 (2) | 1 (1) | 0 (0) | 2 (3)
Dyslexia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 4 (4) | 18 (24) | 2 (3) | 1 (1) | 0 (0) | 8 (11)
Hemianopia homonymous (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 8 (9) | 3 (3) | 3 (3) | 1 (1) | 4 (4)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Muscle spasticity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (9) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual field defect (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Decreased interest (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 2 (2) | 0 (0) | 1 (1) | 4 (4)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Persistent depressive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 14 (16) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 2 (2)
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/62/NCT03150862/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/62/NCT03150862/SAP_001.pdf